CLINICAL TRIAL: NCT03092258
Title: Do we Prepare Patients for Their Digital Legacy? A Survey of Palliative Care Professionals in the West Midlands
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017PAL90
Record Dates: First submitted 2017-03-14; First posted 2017-03-27 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Death
MeSH Terms: conditions — Death | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire to be completed by staff

SUMMARY:
Conduct a questionnaire survey of palliative care professionals including doctors, nurses and social workers currently working within the West Midlands to establish how much the palliative care community in the West Midlands engage in preparing patients for their digital legacy and find out if there is a further education need in this community about digital legacy.

ELIGIBILITY:
Inclusion Criteria:

* Palliative care professionals (medical, nursing and social worker) affiliated to a hospice in the West Midlands.

Exclusion Criteria:

* Medical, nursing or social worker not working in a hospice in the West Midlands.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Palliative care professionals (medical, nursing and social worker) affiliated to a hospice in the West Midlands.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Professionals' behaviour. | 6 weeks
  Questionnaire establishing a baseline measure from which to monitor changes over time in professionals' behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Hazel Coop, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- Compton Hospice, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No